CLINICAL TRIAL: NCT00451191
Title: Intraprostatic Injection of Botulinum Toxin for the Management of Benign Prostatic Hyperplasia: A Randomized Phase II Trial
Brief Title: Botulinum Toxin Injection for the Management of BPH
Acronym: MIST2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIST2; U01DK060817 (NIH); NCT00395525 (obsolete NCT alias)
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; BPH; botulinum toxin; BoNT/A
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): 100 units botulinum toxin type A (BoNT/A)
  Interventions: Drug: botulinum toxin type A (BoNT/A)
- 2 (Active Comparator): 300 units botulinum toxin type A (BoNT/A)
  Interventions: Drug: botulinum toxin type A (BoNT/A)

INTERVENTIONS:
Drug: botulinum toxin type A (BoNT/A) — 100 unit and 300 unit dosages: Dilute each 100 U vial with 1.3 ml of normal saline. Each reconstituted vial is then drawn up into a single syringe with a total of 4 ml = 300 U. The instrument used to inject the botulinum toxin is an ultrasound device with a transrectal ultrasound probe specially designed for prostate biopsies which has a special canal to introduce and direct a needle in to the selected prostatic area.
  Other Names: marketed in the US as BOTOX by Allergan

SUMMARY:
This is a double-blind randomized phase II trial to determine whether two different doses of BoNT/A injection into the prostate gland demonstrate sufficient improvement in the management of lower urinary symptoms due to BPH to warrant more extensive research. Subjects will receive either a 100U or 300U dose. Participation will last 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male at least 50 years of age.
* Voided volume => 125 ml.
* Maximum urinary flow < 15 ml/sec.
* AUA symptom severity score => 8.
* Patient signed informed consent prior to the performance of any study procedures.
* Patient able to complete the study protocol in the opinion of the investigator.

Exclusion Criteria:

* Any prior surgical intervention for BPH.
* Current diagnosis of acute or chronic prostatitis (which may cause LUTS that mimic BPH).
* Overactive bladder without bladder outlet obstruction.
* Enrolled in another treatment trial for any disease within the past 30 days.
* Men interested in future fertility.
* Previous exposure to botulinum toxin.
* On alpha-blocker within the past 48 hours.
* On any 5-alpha-reductase inhibitor within the past month.
* Post void residual > 350 ml.
* On phenylephrine, pseudoephedrine, imipramine, an anticholinergic, or cholinergic medication within the past 2 weeks.
* On estrogen, androgen, any drug producing androgen suppression, or anabolic steroids within the past 4 months.
* Clinically significant renal or hepatic impairment as determined by abnormal creatinine or AST levels (based on local institutional values).
* Serum prostate specific antigen level > 8 ng/ml (Hybritech). For those with a PSA between 4-8 ng/ml, the PSA elevation must be considered to be from a benign cause in the opinion of the PI. This decision can be based on PSA velocity, previous TRUS biopsy, percent free PSA, or other clinical estimations in keeping with sound urologic care.
* Active urinary tract disease or biopsy of the prostate within the past 6 weeks.
* Daily use of a pad or device for incontinence required.
* Episode of unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident (stroke) within the past 6 months.
* On aminoglycosides or any drug that interfere with neuromuscular transmission.
* Eaton-Lambert syndrome, hemophilia, hereditary clotting factors deficiency, or bleeding diathesis.
* Penile prosthesis or artificial urinary sphincter.
* History or current evidence of carcinoma of the prostate or bladder, pelvic radiation or surgery, urethral stricture, or bladder neck obstruction.
* Known primary neurologic conditions such as multiple sclerosis, myasthenia gravis or Parkinson's disease, or other neurological diseases known to affect bladder function.
* Documented bacterial or acute prostatitis within the past year.
* Two documented urinary tract infections of any type in the past year (UTI defined as > 100,000 colonies per ml urine from midstream clean catch or catheterized specimen).
* History of bladder calculi.
* Patients must be off aspirin, NSAIDS, and Coumadin for 7 or more days prior to botulinum toxin injection.
* Cancer that is not considered cured, except basal cell or squamous cell carcinoma of the skin (cured defined as no evidence of cancer within the past 5 years).
* Any serious medical condition likely to impede successful completion of the study, such as certain mental disorders, hypersensitivity to botulinum toxin or anesthetics used in the study, syncope, uncontrolled diabetes.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Bruskewitz, MD, Study Chair — University of Wisconsin, Madison
Locations (7):
- United States (7):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Cornell University, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository https://repository.niddk.nih.gov/studies/mist2/?query=mist
URL: https://repository.niddk.nih.gov/studies/mist2/?query=mist

REFERENCES:
- [Result] Crawford ED, Hirst K, Kusek JW, Donnell RF, Kaplan SA, McVary KT, Mynderse LA, Roehrborn CG, Smith CP, Bruskewitz R. Effects of 100 and 300 units of onabotulinum toxin A on lower urinary tract symptoms of benign prostatic hyperplasia: a phase II randomized clinical trial. J Urol. 2011 Sep;186(3):965-70. doi: 10.1016/j.juro.2011.04.062. Epub 2011 Jul 24. PMID 21791356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the 7 clinical centers (Baylor College of Medicine, Houston TX; Cornell University, New York NY; Mayo Clinic, Rochester MN; Medical College of Wisconsin, Milwaukee WI; Northwestern University, Chicago IL; University of Colorado Denver, Aurora CO; University of Texas Southwestern Medical Center, Dallas TX).
Pre-assignment Details: Screening for eligibility: male, 50+ years old, signed informed consent, no prior surgical treatment for BPH and no prior use of botulinum toxin, appropriate washout period for medical therapy, American Urological Association Symptom Index (AUASI) >=8, voided volume >=125 ml, maximum urinary flow rate <15 ml/sec.
Groups:
- 100 Units Botulinum Toxin Type A; 300 Units Botulinum Toxin Type A: botulinum toxin type A (BoNT/A) : 100 unit and 300 unit dosages: Dilute each 100 U vial with 1.3 ml of normal saline. Each reconstituted vial is then drawn up into a single syringe with a total of 4 ml = 300 U. The instrument used to inject the botulinum toxin is an ultrasound device with a transrectal ultrasound probe specially designed for prostate biopsies which has a special canal to introduce and direct a needle in to the selected prostatic area.
Period: Overall Study
Arm/Group | 100 Units Botulinum Toxin Type A | 300 Units Botulinum Toxin Type A
Started | 68 | 66
Completed | 53 | 55
Not Completed | 15 | 11
Not completed — withdrawal or received alternate tx | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 Units Botulinum Toxin Type A | 300 Units Botulinum Toxin Type A | Total
Number analyzed (Participants) | 68 | 66 | 134
Age, Customized [Number; unit: participants]
  <50 years | 0 | 0 | 0
  >=50 years | 68 | 66 | 134
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 68 | 66 | 134
Region of Enrollment [Number; unit: participants]
  United States | 68 | 66 | 134

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the AUA Symptom Score Index by 30% From Baseline Within the First 12 Weeks After Injection.
Description: The primary outcome was treatment success at 3 months post-treatment, defined as (1) improvement in the AUASI by at least 30% and/or (2) Qmax improvement of more than 30%, each determined from baseline to 3 months after injection. In addition, two safety criteria also had to be met; a dose failed if (1) any reported event was determined to be related to the onabotulinum toxin A injection and was considered life threatening, disabling, or fatal or (2) >=40% of the participants reported a moderate or severe side effect related to the botulinum toxin injection.
Time Frame: 12 weeks
Population: By the last 12-month follow-up visit, 15 men (22%) in the 100 U dose arm and 11 (17%) in the 300 U dose arm had withdrawn due to dissatisfaction with treatment results or continued to attend study follow-up but received additional alternate treatment prior to 12 months.
Measure: Number; unit: participants
Arm/Group | 100 Units Botulinum Toxin Type A | 300 Units Botulinum Toxin Type A
Number analyzed (Participants) | 53 | 55
participants | 46 | 50
Statistical Analysis 1: Comparison: 100 Units Botulinum Toxin Type A vs 300 Units Botulinum Toxin Type A; Simon's optimal two-stage design was applied to determine whether there was sufficient activity at either of the two dose levels to warrant further investigation. Each patient was considered either a successful or failed response. The response rate or proportion of patients treated successfully was examined in two stages. At both stages, the two dose levels were compared to pre-determined critical cut-off values. Sample size was based on significance level α=0.05 and power 90%; Test type: Superiority or Other; p < 0.05, Simon's optimal two-stage design

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse and serious adverse events were collected at scheduled study visits or by participant contact between visits. A standard form was completed.
Arm/Group | 100 Units Botulinum Toxin Type A | 300 Units Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 7/68 | 5/66
Other Adverse Events (participants affected / at risk) | 46/68 | 41/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 Units Botulinum Toxin Type A (N=68) | 300 Units Botulinum Toxin Type A (N=66)
Grade 2 - 4 Serious Adverse Event (General disorders) | 6 (6) | 5 (6) — In 100 U Arm there were 3 SAEs and in 300 U Arm there were 5 SAEs that were not related to study treatment/procedures
Grade 5 Serious Adverse Event (Death) (General disorders) | 1 (1) | 0 (0) — In 100 U Arm, death was not related to study treatment/procedures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 Units Botulinum Toxin Type A (N=68) | 300 Units Botulinum Toxin Type A (N=66)
Grade 1-3 Adverse Event (General disorders) | 46 (116) | 41 (109) — In 100 U Arm there were 64 AEs and in 300 U Arm there were 64 AEs that were not related to study treatment/procedures

LIMITATIONS AND CAVEATS:
First, this study was not designed to compare the effect of onabotulinum toxin A to placebo. Second, we assessed our primary outcome, treatment efficacy, at 3 months post-injection. The long-term safety of this product should also be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No